CLINICAL TRIAL: NCT02065609
Title: Assessment of HER2 Receptors in Breast Carcinoma by Positron Emission Tomography (PET) Using 89 Zr-Trastuzumab
Brief Title: 89ZrTrastuzumab Breast Imaging With Positron Emission Tomography
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Professor of Radiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201307037; R21CA182945 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-19 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 89Zr-Trastuzumab Human Dosimetry and Safety
  Interventions: Drug: 89Zr-Trastuzumab Human Dosimetry and Safety; Drug: HER2 Positive Lesion Detection and Safety
- Cohort 2: Lesion Detection and Safety (Experimental): HER2 Positive Lesion Detection and Safety
  Interventions: Drug: 89Zr-Trastuzumab Human Dosimetry and Safety; Drug: HER2 Positive Lesion Detection and Safety

INTERVENTIONS:
Drug: 89Zr-Trastuzumab Human Dosimetry and Safety — PET Imaging following administration of 89Zr labeled Trastuzumab for calculation of human dosimetry and overall safety
Drug: HER2 Positive Lesion Detection and Safety — Detection of HER2 Positive Breast Cancer with 89Zr Labeled Trastuzumab and PET imaging

SUMMARY:
The main purpose of this study is to see if Positron Emission Tomography (PET-Imaging) with 89Zr labeled trastuzumab can detect trastuzumab (HER2) positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Cohort 1: Her2-positive (defined as 3+) or FISH HER2:CEP17 ratio > 2 biopsy proven breast cancer
* Cohort 2: Her2-positive (defined as 3+) or FISH HER2:CEP17 ratio > 2 OR HER2negative (0 or 1+, 2+ and FISH negative) biopsy-proven breast cancer
* Primary or recurrent/metastatic lesion size ≥ 1.5 cm as determined by imaging studies (ultrasonography, mammography, CT or MRI) or physical examination
* Able to give informed consent
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 89Zr-trastuzumab) is negative
* Patients currently receiving trastuzumab therapy with or without other types of systemic therapy can participate if their disease progresses (development of new lesion(s) or worsening of known lesion(s) based on imaging modalities or physical examination.

Exclusion Criteria:

* Patients with other invasive malignancies, with the exception of non- melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years
* Unable to tolerate 60 min of PET imaging per imaging session

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine @ Barnes-Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study first enrollment occurred in February 2014 and closed to enrollment 31 December 2017. Subjects were recruited from those patients being seen by medical oncology at Siteman Cancer Center. Planned enrollment was 67 participants with a total of 52 subjects enrolled with evaluable data at the end of the grant period.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2: Lesion Detection and Safety
Started | 12 | 40
Completed | 12 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2: Lesion Detection and Safety | Total
Number analyzed (Participants) | 12 | 40 | 52
Age, Customized [Mean (Full Range); unit: years] | 56.9 [29 to 74] | 56 [37 to 78] | 56.5 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 40 | 52
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 39 | 51
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 40 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability After 89Zr-Trastuzumab Administration
Description: Subjects medical record was followed for 30 days following 89Zr-Trastuzumab Administration for AE Assessment with AE being defined as Any unfavorable medical occurrence in a human subject who receives 89Zr-Trastuzumab and PET/CT imaging, including any abnormal sign, symptom, or disease. The event does not necessarily have to be causally related to injection of 89Zr-Trastuzumab or PET/CT imaging to qualify as an adverse event, just temporally related.
Time Frame: 30 Days following 89Zr-Trastuzumab Administration
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2: Lesion Detection and Safety
Number analyzed (Participants) | 12 | 40
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events for the 30 days following 89Zr-Trastuzumab administration
Description: AE assessment was based on the following: Any unfavorable medical occurrence in a human subject who receives 89Zr-Trastuzumab and PET/CT imaging, including any abnormal sign, symptom, or disease. The event does not necessarily have to be causally related to injection of 89Zr-Trastuzumab or PET/CT imaging to qualify as an adverse event, just temporally related. The event of kidney injury and sepsis noted at 30 day follow up was directly related to SOC therapy and not considered study related AE
Arm/Group | Cohort 1 | Cohort 2: Lesion Detection and Safety
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/40
Other Adverse Events (participants affected / at risk) | 1/12 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2: Lesion Detection and Safety (N=40)
non-neutropenic fever (General disorders) | 1 (2) | 0 (0) — One Cohort 1 subject presented with non-neutropenic fever and flu like symptoms 1 day after administration of 89Zr-Trastuzumab and 2 days after receiving standard of care chemotherapy. Subject had similar presentation with prior cycle of SOC therapy
Flu Like Symptoms (General disorders) | 1 (2) | 0 (0) — One Cohort 1 subject presented with non-neutropenic fever and flu like symptoms 1 day after administration of 89Zr-Trastuzumab and 2 days after receiving standard of care chemotherapy. Subject had similar presentation with prior cycle of SOC therapy
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (2) — Cohort 2 subject presented 26 days post administration of 89Zr-Trastuzumab with sepsis and renal injury
Sepsis (Infections and infestations) | 0 (0) | 1 (2) — Cohort 2 subject presented 26 days post administration of 89Zr-Trastuzumab with sepsis and renal injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT02065609/Prot_SAP_ICF_000.pdf